CLINICAL TRIAL: NCT05023668
Title: China Atopic Dermatitis Registry Study: a Chinese Registry Study in Moderate-to-severe Atopic Dermatitis Patients Not Controlled by Topical Therapy
Brief Title: China Atopic Dermatitis Registry Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang jianzhong, Professor and Chairman, Department of Dermatology, Peking University People's Hospital
Other Study IDs: SGZ-2020-12888
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese moderate to severe atopic dermatitis patients not controlled by topical therapy: Chinese moderate to severe atopic dermatitis patients not controlled by topical therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This regestry study is aimed to characterize the medical care and drug treatment under real-life conditions among Chinese patients with moderate to severe Atopic Dermatitis who are not well controlled by topical therapies.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic recurrent inflammatory skin disease, resulting in itchy, red, and skin lesion. A survey conducted in 2014 in 39 tertiary hospitals of 15 provinces in mainland China has shown that the incidence of AD in outpatients (7.8%) has been raised in recent years.

Among topical therapy of AD, corticosteroids are first line therapy. In patients with extensive and severe dermatitis, topical therapy may be insufficient. Such patients may require the addition of either oral corticosteroid or systemic immunosuppressive therapy and even phototherapy. There is no clear recommendation treatment for each kind of patients with different severity yet and there are still huge unmet medical needs for treatment. There is not clear recommendation grade for these therapy in Chinese AD guideline and no published data to demonstrate current treatment situation in real clinical practise.

The goal of clinical registry study is to document the use and effectiveness of therapeutic interventions under real-life conditions. This study will help understand the clinical characteristics, treatment utilization, treatment patterns, as well as disease-related outcomes and cost among AD patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Age≥12;
* AD according to Williams diagnosis criteria (see Appendix 1);
* Moderate to severe AD that inadequately controlled by topical therapy
* Moderate-to-severe: SCORAD score≥25; or
* Inadequately controlled by topic therapies: Determined by physicians.

Exclusion Criteria:

* No.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Chinese moderate-to-severe atopic dermatitis patients who are not controlled by topical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Physician evaluated effectiveness of Atopic Dermatitis therapies in real life | At Month 12
  Physician-reported outcome tool, SCORAD index, will be used to evaluate the objective severity of clinical signs of Atopic Dermatitis .
Patient-reported disease symptoms after Atopic Dermatitis therapies in real life | At Month 12
  Patient Oriented Eczema Measure (POEM) will be used to assess disease symptoms
Patient-reported severity of pruritus after Atopic Dermatitis therapies in real life | At Month 12
  Peak Pruritus Numerical Rating Scale (NRS) will be used to assess severity of pruritus.
Patient-reported disease control after Atopic Dermatitis therapies in real life | At Month 12
  Atopic Dermatitis Control Tool (ADCT) will be used to assess long term disease control.
Patient-reported quality of life after Atopic Dermatitis therapies in real life | At Month 12
  Dermatology Life Quality Index (DLQI) will be used to assess quality of life, and DLQI for children (cDLQL) will be used for adolescence patients.
The Atopic Dermatitis related economic burden | At Month 12
  Economic burden of Atopic Dermatitis will be evaluated using the cost of hospitalizations and outpatient visits associated with Atopic Dermatitis during the past one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu P, Lin B, Shen Y, Lu Y, Li J, Lv D, Yao X, Man X, Fang H, Jiang G, Yu N, Liu D, Zhan S, Zhang J. The ChinaSTAD Chinese Registry in Patients with Moderate-To-Severe Atopic Dermatitis Not Controlled by Topical Therapy: Baseline Characteristics, Disease Burden and Treatment. Dermatol Ther (Heidelb). 2025 Nov;15(11):3377-3389. doi: 10.1007/s13555-025-01540-w. Epub 2025 Sep 19. PMID 40971027